CLINICAL TRIAL: NCT05443984
Title: A Randomized, Double-blind, Parallel, Active-controlled, Non-inferiority, Phase III Multiple Center Clinical Trial to Compare the Efficacy and Safety of JP-1366 20 mg Versus Esomeprazole 40 mg in Patients With Erosive Esophagitis
Brief Title: JP-1366 20mg Versus Esomeprazole 40mg in Patients With Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JP-1366-301
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2022-07

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): JP-1366 20mg + Esomeprazole 40mg(placebo)
  Interventions: Drug: JP-1366 20mg
- Active Comparative Group (Active Comparator): JP-1366 20mg(placebo) + Esomeprazole 40mg
  Interventions: Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: JP-1366 20mg — 1 capsule of JP-1366 20 mg, 1 tablet of esomeprazole placebo (irrespective of meals)
  Arms: Experimental Group
Drug: Esomeprazole 40mg — 1 capsule of JP-1366 placebo, 1 tablet of esomeprazole 40 mg placebo (irrespective of meals)
  Arms: Active Comparative Group

SUMMARY:
To evaluate the efficacy and safety of JP-1366 20 mg compared to esomeprazole 40 mg in patients with erosive esophagitis

ELIGIBILITY:
* Inclusion Criteria: Subjects must satisfy all the following criteria.

  1. Male or female, ≥ 19 years of age at the time of obtaining consent
  2. Subjects who had experienced heartburn and regurgitation within 7 days prior to the screening visit, those whose severity and frequency of symptoms fall under the following (1) or (2)

     ⑴ Subjects who have experienced mild or more severe heartburn or regurgitation at least twice a week

     ⑵ Subjects who have experienced moderate or more severe heartburn or regurgitation at least once a week
  3. Endoscopically confirmed grade A or higher erosive esophagitis as defined by †LosAngeles classification within 15 days, prior to randomization
  4. Subjects who fully understand this study and voluntarily signed on the informed consent form
* Exclusion Criteria: Subjects may not satisfy any of the following criteria.

  1. Subjects who can't undergo endoscopy
  2. Medical History

     º Subjects who have warning symptoms of the malignant gastrointestinal tract such as odynophagia, severe dysphagia, bleeding, weight loss, anemia, or bloody stool. (except negative result for malignancy by endoscopy)

     º Subjects with eosinophilic esophagitis (except negative result by esophageal biopsy)

     º Subjects who have esophageal stenosis, gastroesophageal varices, Barrett's esophagus, active gastric ulcer, gastrointestinal bleeding, or malignant tumor confirmed by EGD

     º Zollinger-Ellison syndrome patients

     º Subjects diagnosed with primary esophageal motility disorder, irritable bowel syndrome (IBS), inflammatory bowel disease (IBD), or suspected with IBS in the last 3 months and with a current history of the disease including pancreatitis

     º Subjects who have a history of gastric acid suppression surgery, gastrointestinal or esophageal surgery (except appendectomy, cholecystectomy, polypectomy)

     º Subjects with a history of clinically significant hepatic, renal, cardiovascular, respiratory, endocrine, urinary, neuro-psychiatric, hemato-oncologic disorder

     º Subjects who have a history of malignant tumor in 5 years at the time of screening. However, excluding subjects with malignant gastrointestinal cancer regardless of the period.
  3. Laboratory Test

     Screening laboratory test showing any of the following abnormal laboratory results:

     º ALT or AST > 2.0 x ULN

     º ALP or GGT > 2.0 x ULN

     º Total bilirubin > 2.0 x ULN

     º eGFR<70 mL/min/1.73 m2 (CKD-EPI formula)

     º Positive result for Serological test (HBsAg, HCV Ab, HIV Ab, Syphilis reagin test)

     º Clinically significant ECG abnormalities
  4. Allergy and drug hypersensitivity

     º Known hypersensitivity to the active ingredient or excipients of the investigational product

     º Clinically significant allergies (except mild allergic rhinitis) or hypersensitivity history to drugs. (Aspirin, antibiotics, etc.)
  5. Prohibited medication and therapy

     º Subjects who take gastric acid suppressant like P-CAB, PPI within 2weeks prior to EGD of screening procedure

     º Subjects who take medication (antacids, prokinetics, H2RA, etc.) related to reflux esophagitis more than 2times within 1week prior to EGD of screening procedure

     º Subjects who need to take medication (aspirin, NSAIDs, etc.) that may cause an ulcer, during the study period

     º Subjects who are on or need to be on the medications which categorized as contraindicated in this clinical trial.

     However, subjects who are on the contraindicated medications can participate in the trial after the washout period of 2 weeks. If five times of the half-life of the contraindicated medications exceeds 2 weeks, the washout period will be set as five times of the half-life.
  6. Pregnant and lactating women
  7. Contraception Subjects who do not agree to use medically acceptable methods of contraception during the period study
  8. Subjects with clinically significant psychiatric disorder and a history with a drug and alcohol abuse.
  9. Subjects who are judged unsuitable to participate in the study in the opinion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
The cumulative healing rate of mucosal break at 8-week after the investigational product administration (%) | Week 8
  The proportion of subjects with remission on endoscopy at 8-week

SECONDARY OUTCOMES:
Healing rate of mucosal break at the 4-week after the investigational product administration | Week 4
  The proportion of subjects whose mucosal breaks are healed on the 4-week endoscopy
Healing rate of mucosal break evaluated by an independent evaluator at the 4-week after the investigational product administration | Week 4
The cumulative Healing rate of mucosal break evaluated by an independent evaluator at the 8-week after the investigational product administration | Week 8
Symptom assessment according to the RDQ questionnaire | Week 4 and 8
Gastro-esophageal symptoms assessment through subject diary at 4, 8 weeks | within 24hours after IP administration, during 7days after IP administration, Week 4 and 8
Change from baseline in the total score of GERD-HRQL at 4, 8-week and cumulative changes in quality of life at 8week | Week 4 and 8

OTHER OUTCOMES:
Exploratory variables | Week 4 and 8
  Healing rate of mucosal break according to H.pylori infection

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center and 26 hospitals, Seoul, South Korea

REFERENCES:
- [Derived] Oh JH, Kim HS, Cheung DY, Lee HL, Lee DH, Kim GH, Choi SC, Cho YK, Chung WC, Kim JW, Yu E, Kwon H, Kim J, Kim J, Jung HY. Randomized, Double-Blind, Active-Controlled Phase 3 Study to Evaluate Efficacy and Safety of Zastaprazan Compared With Esomeprazole in Erosive Esophagitis. Am J Gastroenterol. 2025 Feb 1;120(2):353-361. doi: 10.14309/ajg.0000000000002929. Epub 2024 Jul 3. PMID 38976448